CLINICAL TRIAL: NCT05325710
Title: Assessment of Personalized Follow-up in Prevention of Type 2 Diabetes
Acronym: Proxipart
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-A00375-36
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-03

CONDITIONS: Diabete Type 2
Keywords: diabete type 2; preventive approach
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Compare a group of patient with study-nurse specific regular follow-up versus standard follow-up in France
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TD2 standard (Active Comparator): Standard TD2 follow-up
  Interventions: Behavioral: Study nurse intervention
- TD2+ study Nurse (Experimental): Specific study nurse follow-up every 4 months in addition of standard FU.
  Interventions: Behavioral: Study nurse intervention

INTERVENTIONS:
Behavioral: Study nurse intervention — Contact everay 4 months with a dedicated study nurse

SUMMARY:
In France, the overall prevalence of diabetes was estimated at 5% of population in 2016, type 2 diabetes (T2DM) corresponding to 90% of cases. However, this figure is greatly underestimated,since it does not take into account people who are untreated or not diagnosed. However,it is estimated that 20 to 30% of adults with diabetes do not are not diagnosed. Conclusions presented during the annual meeting of the european Association for the Study of diabetes (EASD-Berlin) from 2019 suggest that signs precursors of the disease would be present up to 20 years before the diagnosis.

The Diagnosis is usually made around 40-50 years. The main factor of risk of T2D is the lifestyle, in particular a diet too rich for a too sedentary daily life.

From a medico-economic point of view, chronic pathologies (including diabetes) account for 60% of insurance expenditure illness even though they concern 35% of insured persons, i.e. 20 million patients. The average annual repayment of a type 2 diabetic patient is 4890 euros.

This study is part of this context as the starting point a reflection on a different, coordinated management, to know a preventive rather than a curative approach.

DETAILED DESCRIPTION:
In France, the overall prevalence of diabetes was estimated at 5% of population in 2016, type 2 diabetes (T2DM) corresponding to 90% of cases. However, this figure is greatly underestimated. since it does not take into account people who are untreated or not diagnosed. However, given the silent nature of the disease, it is estimated that 20 to 30% of adults with diabetes do not are not diagnosed. This share decreases with age, falling to 13% among 55-74 year olds. Conclusions presented during the annual meeting of the european Association for the Study of diabetes (EASD-Berlin) from 2019 suggest that signs precursors of the disease would be present up to 20 years before the diagnosis.

Type 2 diabetes, or non-insulin dependent diabetes, is a metabolic disease characterized by a chronic excess of sugar in the blood, affecting both men and women. the Diagnosis is usually made around 40-50 years. The main factor of risk of T2D is the lifestyle, in particular a diet too rich for a too sedentary daily life. The direct consequences are an increase in obesity hich is itself a major risk factor for the development of T2D. Among the risk factors, we also find hyperlipidemia, high blood pressure, high blood sugar fasting, stress, smoking, heredity, family history of diabetes, or gestational diabetes.

From a medico-economic point of view, chronic pathologies (including diabetes) account for 60% of insurance expenditure illness even though they concern 35% of insured persons, i.e. 20 million patients. The average annual repayment of a type 2 diabetic patient is 4890 euros.This study is part of this context as the starting point a reflection on a different, coordinated management, to know a preventive rather than a curative approach.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over the age of 18
* Patient with a FINDRISC score ≥10 points
* Beneficiary of a French health insurance system
* Patient having been informed and having given their consent free, enlightened and written

Exclusion Criteria:

* Patient over 75 years old
* Patient already diagnosed with type 2 diabetes
* Patient whose physical and/or psychological health is severely impaired, which according to the investigator may affect the compliance of the study participant.
* Patient participating in another research
* Patient in period of exclusion from another research always in progress at the time of inclusion.
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by court order or administration.
* Pregnant, breastfeeding or parturient women.
* Patient hospitalized without consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2022-03-20 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
FINDRISC score | 5 years
  FINDRISC is a prediction tool to identify patients at risk of developing diabetes without biological analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Aguiléra, Biarritz, Aquitaine, France

IPD SHARING:
Plan to Share IPD: Undecided